CLINICAL TRIAL: NCT02362243
Title: Worksite Exercise Interventions for Low Back Injury Prevention in Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Federal Emergency Management Agency (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EMW-2013-FP-00723
Record Dates: First submitted 2015-02-06; First posted 2015-02-12 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Low Back Pain
Keywords: low back pain; low back injury; firefighter; prevention; physical fitness; exercise training; worksite; web-based
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (Placebo Comparator): Participants in the control arm will complete the placebo comparator intervention.
  Interventions: Other: Placebo Comparator
- Supervised Exercise Group (Experimental): Participants in the supervised exercise intervention arm will perform the experimental intervention under direct 1-on-1 supervision of an exercise specialist.
  Interventions: Other: Experimental Intervention
- Web-based Exercise Group (Experimental): Participants in the web-based exercise intervention arm will perform the experimental intervention with use of a web-based exercise system for exercise instruction and guidance, and without direct 1-on-1 on-site supervision.
  Interventions: Other: Experimental Intervention

INTERVENTIONS:
Other: Experimental Intervention — Participants will perform the back and core exercises that were tested in our previous firefighter study (Mayer, 2015), in addition to their usual physical fitness routine. All participants at a given fire station will receive the same intervention and all interventions will be completed at the fire station. Participants will perform 2 exercise sessions each week (each time they are on duty) throughout the study's 12-month duration. The back and core exercise program consists of 1 set of 5 exercises - 4 core exercises on a floor mat and 1 back extension exercise on a variable angle Roman chair - which will take approximately 10 minutes to complete for each session (Mayer, 2015).
  Arms: Supervised Exercise Group; Web-based Exercise Group
Other: Placebo Comparator — Participants will receive a 45-60 minute, one-time educational session, which will be delivered to delivered by an exercise specialist in a 1-on-1 format while the participant is on-duty at the fire station, in addition to their usual physical fitness routine. Content for the educational session on evidence-based guidelines for exercise, physical fitness, and general physical activity will be derived from the American College of Sports Medicine (ACSM) Position Stand - Quantity and Quality of Exercise for Developing and Maintaining Cardiorespiratory, Musculoskeletal, and Neuromotor Fitness in Apparently Healthy Adults: Guidance for Prescribing Exercise (Garber, 2011).
  Arms: Control Group

SUMMARY:
Purpose and Aims: The purpose of this study is to assess the clinical effectiveness of back and core exercise interventions for low back injury prevention in firefighters. Aim 1. Compare the effectiveness of 2 worksite exercise interventions (supervised, web-based) relative to control to reduce lost work days related to low back injury and illness in firefighters.

Relevance: Low back injury is one of the most common and disabling disorders in firefighters. Thus, novel interventions are needed to counteract the adverse consequences of this disorder and its impact on firefighter safety.

Methods: A cluster randomized controlled trial will be conducted in career, full active duty firefighters (n = 345) who will be randomly assigned (by fire station) to 1 of 3 intervention groups - 1) supervised exercise (n = 115), 2) web-based exercise (n = 115), or 3) control (n = 115). Participants in the supervised and web-based exercise groups will perform back and core exercises previously tested in our recent FEMA-funded grant (EMW-2009-FP-00418), twice per week for 12 months while on duty, in addition to their usual physical fitness routine - The supervised group will perform exercise under direct supervision of certified exercise specialists, and the web-based group will utilize a web-based exercise system. The control group will not perform back and core exercises, but will continue their usual physical fitness routine and receive brief education on general exercise and physical activity principles. Outcome measures include low back injury and illness data obtained and cross-checked from various sources, other standard clinical outcome measures for low back pain and disability, and validated physical fitness tests.

Anticipated Outcomes: We hypothesize that the supervised and web-based interventions will reduce lost work days related to low back injury and illness by 40% compared with control. Assuming positive results, this study will deliver an evidence-based exercise intervention for low back injury prevention specifically designed for firefighters and assessed in a full-scale randomized controlled trial.

DETAILED DESCRIPTION:
Low back injury is one of the most common and disabling disorders in firefighters (IAFF, 2008). Thus, novel interventions are needed to counteract the adverse consequences of this disorder and its impact on firefighter safety. Our long-term research objective is to develop and test interventions to reduce the incidence, morbidity, economic, and other adverse consequences of low back injury and illness in firefighters. Our previous studies funded by the FEMA Assistance to Firefighters Grant Program demonstrated that: 1) a relationship exists between poor back muscular endurance and increased prevalence of low back pain in firefighters (Verna, 2010); and 2) a worksite intervention including back and core exercise training is safe and effective in improving back and core muscular endurance in firefighters (Mayer, 2015). The purpose of the current study, which builds upon our previous work, is to assess the clinical effectiveness of back and core exercise interventions for low back injury prevention in firefighters.

Specific Aims (Purpose) Aim 1. Compare the effectiveness of 2 worksite exercise interventions (supervised, web-based) relative to control to reduce lost work days related to low back injury and illness in firefighters.

Hypotheses: Primary - The supervised exercise intervention will reduce the number of lost work days related to low back injury and illness over the 12-month intervention period by 40% compared with control. Secondary - The web-based exercise intervention will reduce the number of lost work days related to low back injury and illness over the 12-month intervention period by 40% compared with control. No difference between the supervised and web-based exercise interventions in lost work days will be observed.

To test the hypotheses, a 3-arm, cluster randomized controlled trial will be conducted in career, full active duty firefighters from 76 stations of 3 fire rescue departments in the Tampa Bay region of Florida. Firefighters (n = 345) will be randomly assigned (by fire station) to 1 of 3 exercise intervention groups - 1) supervised, (n = 115), 2) web-based (n = 115), or 3) control (n = 115). Participants in the supervised and web-based exercise groups will perform back and core exercises previously tested in our recent FEMA-funded grant (EMW-2009-FP-00418), twice per week for 12 months, in addition to their usual physical fitness routine. All participants at a given fire station will receive the same intervention and interventions will be completed during normal shift hours at the fire station. The supervised group will perform back and core exercises with on-site, 1-on-1, direct supervision by certified exercise specialists (e.g. peer fitness trainers from the partner fire departments) for each exercise session using an identical strategy as our previous study. The web-based group will be provided an interactive web-based delivery, guidance, and monitoring system for back and core exercises using technology developed by our group and partners, along with remote interaction with and guidance from exercise specialists. The control group will not perform back and core exercises, but will continue their usual physical fitness routine and receive brief education on general exercise and physical activity principles.

Outcome measures to test these hypotheses include low back injury and illness data obtained and cross-checked from various sources, including administrative data (primary outcome), such as reports from the fire departments and workers' compensation data, and participant self-reported questionnaires in accordance with departmental, Occupational Safety and Health Administration (OSHA), and fire service standards. Numerous other clinically relevant measures for low back pain injury and illness, comorbidities, risk factors, and prognosis will also be collected and analyzed, such as incidence, frequency, severity, chronicity/duration, physical function, psychological measures (e.g. fear avoidance), back and core muscular endurance, body mass index, Functional Movement Screen, physical activity and exercise measures, and cost-effectiveness. In order to inform implementation efforts throughout the fire service, we will conduct a health economic analysis, such as cost effectiveness, and collect data to gain a better understanding of the context for implementation of the exercise interventions.

Potential impact on firefighter health and safety. The proposed study will provide pivotal evidence for dissemination and implementation throughout the fire service. Assuming positive results, this study will deliver an evidence-based exercise intervention for low back injury prevention specifically for firefighters and assessed in a full-scale randomized controlled trial.. The innovative, efficient, and effective exercise intervention will reduce the adverse consequences of low back injury and illness in firefighters, and will be ready for national implementation throughout the fire service for fire departments with similar characteristics as those tested. If successfully implemented, this low back injury prevention program will improve firefighter safety and health in order to enhance resilience and preparedness, so they can more effectively carry out their duties to protect the community. Further, this low back injury prevention program will help improve off-duty and long-term quality of life for firefighters.

Unique contribution to body of knowledge. Knowledge gaps exist in evidence-based approaches for low back injury prevention in firefighters, particularly regarding interventions for clinical effectiveness, costs, and implementation. The proposed study will assess such an intervention, and is responsive to 4 health and wellness priorities of the 2011 National Fire Service Research Agenda (NFFF, 2011): 1.0: Health and disease related to firefighter wellness and fitness; 3.0: Implementation / translational research; 7.0: Optimization of performance and reducing risk; and 8.0: Cost effectiveness of health and safety systems.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Full duty, regular service, career firefighter housed at a standard fire station from Hillsborough County Fire Rescue, St. Petersburg Fire & Rescue, or Tampa Fire Rescue.

Exclusion Criteria:

* Current workers' compensation or personal injury case or litigation
* Research personnel (e.g. firefighter peer fitness trainers).
* Participant in the exercise intervention group of our previous FEMA-funded study (EMW-2009-FP-00418).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2016-03; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Mean number of lost work days per participant over a 12-month period due to work-related injury or illness in the low back region | 12 months

SECONDARY OUTCOMES:
Incidence rate of lost work days due to work-related injury or illness in the low back region | 12 months
Time to event of an episode of lost work days due to work-related injury or illness in the low back region | 12 months
Number of episodes of lost work days due to work-related injury or illness in the low back region | 12 months

OTHER OUTCOMES:
Onset of low back injury and illness | Baseline, monthly; upon occurrence
Severity of low back injury and illness | Baseline, monthly; upon occurrence
Mechanism of low back injury and illness | Baseline, monthly; upon occurrence
Healthcare utilization of low back injury and illness | 12 months
Frequency of low back injury and illness | Baseline, monthly; upon occurrence
Current exercise / physical activity habits | Baseline, 3/6/9/12 months
  International Physical Activity Questionnaire
Health-related quality of life | Baseline, 3/6/9/12 months
  SF-12 questionnaire
Low back disability and physical function | Baseline, 3/6/9/12 months
  Oswestry Disability Index
Back beliefs | Baseline, 3/6/9/12 months
  Back Beliefs Questionnaire
Back muscular endurance | Baseline, 12 months
  Modified Biering-Sorensen Isometric Back Endurance Test
Core muscular endurance | Baseline, 12 months
  Isometric Prone Plank Test
Functional movement quality | Baseline, 12 months
  Functional Movement Screen
Participation rate | Baseline, 3/6/9/12 months
  Number of individuals responding to study recruitment, completing initial screening, subsequent screening, enrolling, and providing data at study endpoints
Adherence to exercise intervention | 3/6/9/12 months
  1. Rate: percentage of prescribed exercise sessions completed
  2. Adherence to exercise progression protocol
Satisfaction with outcome | 12 months
  Satisfaction with Outcome Questionnaire
Barriers and facilitators to interventions | 12 months
  Questionnaire
Cost of intervention | 12 months
  Health economic evaluation using various measures
Stages of change | baseline, 12 months
  Stages of Change Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: John M Mayer, DC, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined.

REFERENCES:
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Mayer JM, Quillen WS, Verna JL, Chen R, Lunseth P, Dagenais S. Impact of a supervised worksite exercise program on back and core muscular endurance in firefighters. Am J Health Promot. 2015 Jan-Feb;29(3):165-72. doi: 10.4278/ajhp.130228-QUAN-89. PMID 24524384
- [Derived] Dagenais S, Hayflinger DC, Mayer JM. Economic Evaluation of an Extended Telehealth Worksite Exercise Intervention to Reduce Lost Work Time from Low Back Pain in Career Firefighters. J Occup Rehabil. 2021 Jun;31(2):431-443. doi: 10.1007/s10926-020-09933-8. Epub 2021 Jan 4. PMID 33394268